CLINICAL TRIAL: NCT06268535
Title: Identification of Anticancer Drugs Associated With Cancer Therapy-related Cardiac Dysfunction: a WHO Pharmacovigilance Database
Brief Title: Identification of Anticancer Drugs Associated With Cancer Therapy-related Cardiac Dysfunction: a Pharmacovigilance Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CaenUH_DL_1
Record Dates: First submitted 2023-11-27; First posted 2024-02-20 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Cancer, Therapy-Related
MeSH Terms: conditions — Heart Failure; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cancer therapy with FDA and/or European Medicines Agency approval on the 30th September 2023 — Disproportionality analysis studying the association between cancer therapy with FDA and/or European Medicines Agency approval on the 30th September 2023 and heart failure or cardiac dysfunction in the World Health Organization pharmacovigilance database.

SUMMARY:
Therapeutic advances have significantly improved the survival of patients with cancer. However, these novel therapies are associated with a concomitant increase in the prevalence of toxicity, including cardiovascular complications of cancer therapy.

Among these adverse drug reactions, heart failure and, more generally, cancer therapy-related cardiac dysfunction are the most concerning cardiovascular complications of cancer therapy, carrying a high morbidity burden and an elevated risk of death.

Patients with both heart failure and cancer have a worse prognosis when compared with heart failure patients with no history of cancer. It is therefore crucial to enhance the identification of patients at a higher risk of cancer therapy-related cardiac dysfunction both before and during treatment, especially when utilizing cancer therapies with known potential cardiovascular adverse drug reactions.

The explosion of new anticancer drugs has led to the potential association of these therapies with cardiac dysfunction.

Using VigiBase, the World Health Organization's (WHO) global pharmacovigilance database, the investigators aimed to assess the relationship between cancer therapy-related cardiac dysfunction and the administration of anti-cancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 29/02/2024
* Patients treated with FDA and/or EMA approved cancer therapies (approval the 30th September 2023).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patients in the World Health Organization (WHO) database of individual safety case reports to 29/02/2024 included with at least one anticander drug.
Sampling Method: Non-Probability Sample
Enrollment: 36580288 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Disproportionality individual case data analysis between heart failure of cardiac dysfunction and cancer therapies | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2024
  A disproportionality analysis is carried out using stepwise selection procedure and taking into account confounding factors (factors known to promote heart failure or cardiac dysfunction).

SECONDARY OUTCOMES:
Description of the population of patients having a heart failure of cardiac dysfunction event with cancer therapies | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2024
  The investigators describe the profile of cases of heart failure of cardiac dysfunction among cancer therapies associated with heart failure or cardiac dysfunction in the main analysis. We particularly focused on factors known to promote heart failure.
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2024
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Legallois D, Da Silva A, Alexandre J, Milliez P, Sabatier R, Blanchart K, Plane AF, Font J, Chretien B, Dolladille C. Identification of anticancer drugs associated to cancer therapy-related cardiac dysfunction: a VigiBase(R) disproportionality analysis. Eur Heart J Cardiovasc Pharmacother. 2025 Aug 12;11(5):459-468. doi: 10.1093/ehjcvp/pvaf027. PMID 40272201